CLINICAL TRIAL: NCT04538820
Title: Dexamethasone Dose for Postoperative Nausea and Vomiting Prophylaxis in Obese Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Bahar SAKIZCI UYAR, medical doctor, Diskapi Yildirim Beyazit Education and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 92/07
Record Dates: First submitted 2020-08-13; First posted 2020-09-04 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Nausea and Vomiting
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (Active Comparator): patients with BMI=18.5-24.9 kg/m2 will be received 4 mg dexamethasone at induction of anesthesia for postoperative nausea and vomiting prophylaxis.
  Interventions: Drug: Dexamethasone 4 mg IV-control
- 4 mg (Active Comparator): patients with BMI>30 kg/m2 will be received 4 mg dexamethasone at induction of anesthesia for postoperative nausea and vomiting prophylaxis.
  Interventions: Drug: Dexamethasone 4 mg IV
- 8 mg (Active Comparator): patients with BMI>30 kg/m2 will be received 8 mg dexamethasone at induction of anesthesia for postoperative nausea and vomiting prophylaxis.
  Interventions: Drug: Dexamethasone 8 mg IV

INTERVENTIONS:
Drug: Dexamethasone 4 mg IV-control — dexamethasone 4 mg will be administered at induction of anesthesia for postoperative nausea and vomiting proflaxis to normal weight patients.
  Arms: control
Drug: Dexamethasone 4 mg IV — dexamethasone 4 mg will be administered at induction of anesthesia for postoperative nausea and vomiting proflaxis to obese patients
  Arms: 4 mg
Drug: Dexamethasone 8 mg IV — dexamethasone 8 mg will be administered at induction of anesthesia for postoperative nausea and vomiting proflaxis to obese patients
  Arms: 8 mg

SUMMARY:
compare the effectiveness of different doses of dexamethasone used for postoperative nausea and vomiting prophylaxis in obese patients and in normal weight patients.

DETAILED DESCRIPTION:
compare the effectiveness of different doses of dexamethasone used for postoperative nausea and vomiting prophylaxis in obese patients.

compare the effectiveness of dexamethasone given in 4 mg and 8 mg doses in obese patients with 4 mg doses of dexamethasone in normal weight patients.

4 mg iv dexamethasone will be administered to normal weight patients at induction of anesthesia. This group will be classified as the control group. In obese patients (BMI>30 kg/m2), one group will receive 4 mg dexamethasone and other group will receive 8 mg dexamethasone at induction.

Patients will receive general anesthesia with volatile anesthetics and tramadol will be administered IV at the end of surgery.

Postoperative nausea and vomiting, postoperative pain, blood glucose, wound infection, time to oral intake, hospital stay will be compared.

ELIGIBILITY:
Inclusion Criteria:

High risk patients for postoperative nausea and vomiting:

* Female
* No smoking
* BMI =18.5-24.9 for control group
* BMI >30 for other groups
* undergo laparoscopic cholecystectomy

Exclusion Criteria:

* Diabetes mellitus

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
postoperative nausea and vomiting (PONV) | PONV scores wİll be record during the ﬁrst 24 hours
  The primary outcome is the overall incidence of PONV during the ﬁrst 24 h, deﬁned as any episode of vomiting or nausea.Nausea will be measured using an 11-point verbal rating scale (VRS) running from 0 (no nausea) to 10 (the worst nausea imaginable). We will deﬁne severe PONV as nausea with a score of at least 4 on the VRS, or vomiting.

SECONDARY OUTCOMES:
postoperative pain: 11-point VRS | Pain will be assessed during the ﬁrst 24 hours
  Pain intensity will be measured using a simple 11-point VRS running from 0 (no pain) to 10 (unbearable pain), at rest and on mobilisation (asking the patient to cough).
oral intake | during the ﬁrst 24 hours
  patients will be asked first oral fluid intake time charge criteria.
blood glucose | at 6 and 10 hours after administration of dexamethasone
  Fingerprick capillary blood glucose concentrations will be measured
Length of Hospital Stay | during the ﬁrst 24 hours
  the time will be recorded when patients are discharged home
wound infection | postoperative 30th day
  Patients will be telephone on the 30th postoperative day and questioned in terms of wound infection

CONTACTS AND LOCATIONS:
Locations (1):
- DiskapiYBERH, Ankara, Turkey (Türkiye)